CLINICAL TRIAL: NCT07318831
Title: A Phase II Trial of Chidamide Combined With Dinutuximab Beta, Irinotecan, and Temozolomide for Refractory or Relapsed Neuroblastoma in Children
Brief Title: Phase II Study of Chidamide-Dinutuximab Beta-Irinotecan-Temozolomide for Refractory/Relapsed Neuroblastoma in Children
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251314
Record Dates: First submitted 2025-12-14; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma (NB); Neuroblastoma in Children
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental)
  Interventions: Drug: Chidamide Combined with Dinutuximab Beta, Irinotecan, and Temozolomide

INTERVENTIONS:
Drug: Chidamide Combined with Dinutuximab Beta, Irinotecan, and Temozolomide — Chidamide (C): 5 mg/10 kg (maximum single dose: 30 mg), administered twice per week. The medication follows a schedule of two weeks on treatment followed by one week off. Specifically, it is taken orally on Days 0, 3, 7, and 10 of each three-week cycle. Chidamide is initiated one day before the start of chemotherapy.

SUMMARY:
This is a Phase II clinical trial investigating the effectiveness and safety of a four-drug combination-Chidamide, Dinutuximab Beta, Irinotecan, and Temozolomide-for children with relapsed or refractory neuroblastoma. The primary goal is to evaluate how well this regimen works to control the cancer, while the secondary goal is to closely monitor its safety and side effects in these young patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically diagnosed neuroblastoma, defined according to the International Neuroblastoma Risk Group (INRG) classification system or the Chinese expert consensus/guideline for pediatric neuroblastoma.
2. Patients with relapsed or refractory neuroblastoma. Relapsed: any patient with recurrent neuroblastoma. Refractory: patients showing an inadequate response (partial response, minor response, or stable disease) to prior therapy, leading to progression.
3. Prior treatment with epigenetic drugs (e.g., HDAC inhibitors, DNA methylation inhibitors) or GD2 monoclonal antibodies does not affect eligibility for this study.
4. Presence of evaluable disease.
5. Performance Status: Lansky score ≥50%, Karnofsky score ≥50%, or ECOG score ≤3.
6. Life expectancy ≥12 weeks.
7. Bone marrow function: Without bone marrow disease: Platelets ≥75×10⁹/L, Absolute Neutrophil Count (ANC) ≥0.75×10⁹/L, Hemoglobin ≥8 g/dL (transfusion allowed). With bone marrow disease: Platelets ≥50×10⁹/L, ANC ≥0.5×10⁹/L, Hemoglobin ≥8 g/dL (transfusion allowed).
8. Renal function: No clinically significant proteinuria (morning urine dipstick <2+). If proteinuria ≥2+ is detected, the protein-to-creatinine (Pr/Cr) ratio must be <0.5 or 24-hour protein excretion must be <0.5 g.
9. Serum creatinine ≤1.5 × ULN; if higher, the calculated glomerular filtration rate (by radioisotope method) must be ≥60 mL/min/1.73 m².
10. Hepatic function: AST or ALT ≤2.5 × ULN and total bilirubin ≤1.5 × ULN. In the presence of liver metastases: AST or ALT ≤5 × ULN and total bilirubin ≤2.5 × ULN.
11. Cardiac function: Left ventricular shortening fraction ≥29% on echocardiogram.
12. Coagulation: For patients not on anticoagulation therapy: INR ≤1.5 and APTT ≤1.5 × ULN. Anticoagulation is allowed if INR or APTT is within the therapeutic range (per institutional standards) and the patient has been on a stable dose for at least two weeks prior to study enrollment.
13. Oxygen saturation >94% on room air.
14. Ability to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patients with CTCAE v5.0 Grade 3 or higher toxicities involving hearing impairment, hematologic disorders, hepatic, or renal diseases.
2. Patients with CTCAE v5.0 Grade 2 or higher neurotoxicity.
3. Major surgical procedure within 14 days prior to the first dose of the study drug.
4. Severe infection (requiring IV antibiotics, antifungals, or antivirals) within one week prior to treatment, or unexplained fever >38.5°C during screening or before the first dose.
5. Congenital or acquired immunodeficiency, or active infectious diseases such as HIV or active hepatitis (with transaminase levels not meeting inclusion criteria; HBV DNA ≥1000 IU/mL; HCV RNA ≥1000 IU/mL). Chronic HBV carriers with HBV DNA <2000 IU/mL may be enrolled if they receive concurrent antiviral therapy during the trial.
6. Any concomitant condition that, in the investigator's judgment, seriously jeopardizes patient safety, may confound the study results, or could impede the patient's completion of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | From enrollment to the end of treatment at 10 weeks

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From enrollment to the end of treatment at 10 weeks
Event-Free Survival(EFS) | From enrollment to the end of treatment at 10 weeks
Duration of Response(DOR) | From enrollment to the end of treatment at 10 weeks
Overall Survival (OS) | From enrollment to the end of treatment at 10 weeks

IPD SHARING:
Plan to Share IPD: Undecided